CLINICAL TRIAL: NCT01587105
Title: Improving Care for Children With Complex Needs (I3CN) Study
Brief Title: Improving Care for Children With Complex Needs
Acronym: I3CN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Rita Mangione-Smith, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CCMS
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Results first posted 2017-02-20 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Medically Complex Children; Care Coordination; Case Manager; Care Manager; Collaborative Care; Disease Management; Patient Care Team or Organization; Managed Care; Children With Chronic Conditions; Children With Special Health Care Needs; Shared Care Plan; Patient Care Plan; Health Care and Resource Utilization; Adherence to Care; Functional Status and Productivity; Health Related Quality of Life; Satisfaction With Care; Care Coordinator; Family Experience of Care; Quality Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Usual Care Group
- Comprehensive Care Management Service (Experimental): Care Coordination through the Comprehensive Care Management Service at Seattle Children's Hospital
  Interventions: Behavioral: Comprehensive Case Management Service

INTERVENTIONS:
Behavioral: Comprehensive Case Management Service — When a child enrolls in the CCM program, the child's parent will work together with the CCM team at Seattle Children's to develop a shared care plan for their child. This plan will include all of the child's routine health care needs and information about what to do when the child gets sick. The parent will also have 24 hour access to an on-call CCM nurse.
  Arms: Comprehensive Care Management Service

SUMMARY:
Seattle Children's Hospital (SCH), in collaboration with several health plans and Washington State Department of Social and Health Services developed the Comprehensive Case Management (CCM) program with the goal to reduce costs of care for medically complex children cared for at SCH as well as improve their health status and the quality of care they receive. The CCM program aims to develop and facilitate a reliable and standardized process that empowers the child's primary care provider and provides him/her with the resources s/he needs to avoid unnecessary emergency department visits and admissions. Our study will include children who had a hospitalization or emergency department visit at Seattle Children's between 2009-2012 and, at that time, had multiple active chronic medical issues but had no specialty service at Seattle Children's to help their primary care providers manage them.

DETAILED DESCRIPTION:
Children with complex health care needs often lack a comprehensive care plan and access to case management. They are at risk for frequent and prolonged hospitalizations, fragmented care, parental stress/burnout and unsafe care. To address this issue, Seattle Children's Hospital developed the Comprehensive Case Management (CCM) program, which includes access to a special clinic at Seattle Children's with case managers and a health care team that works with parents and community physicians to create care plans for children with complex needs.

The investigators goal is to evaluate whether children who participate in the CCM program have better parent reported access to needed care, timeliness of receiving needed services, more coordinated care, improved health status, and higher parent satisfaction with care compared to children who receive care outside the CCM program. In addition, the investigators will examine whether these children experience decreased annual costs of care, emergency department visits, hospital admissions, and hospital lengths of stay compared to children receiving care outside the program. The investigators also want to understand whether community physicians who have patients enrolled in the CCM program are more satisfied with caring for children with complex medical needs than physicians caring for these children outside the program.

The investigators plan to enroll 650 parents of eligible children into the I3CN study. Three hundred twenty five of these parents will have children enrolled in the CCM program and 325 will have children who continue to receive usual care. Enrolled parents complete a survey every 6 months during the study (5 surveys over 2 ½ years) in order to assess study outcomes including parent perceived. Parent participation in the study will be completed 2 ½ years after enrollment.

When a child enrolls in the CCM program, the child's parent will work together with the CCM team at Seattle Children's to develop a shared care plan for their child. The CCM team includes physicians, nurse practitioners, social workers, nutritionists, and nurse case managers. This plan will include all of the child's routine health care needs in addition to information about what to do when the child gets sick. Community providers will also be asked to review and provide input on the shared care plan. Once the shared care plan is in place, the parent, primary care provider (PCP), and the CCM clinic will follow the standardized processes established by the program and the shared care plan when the child becomes ill.

During the course of the 2 ½ year study, the investigators will analyze our outcomes of interest every 6 months. If the investigators find that children in the CCM the program are experiencing significantly better outcomes than children receiving care outside the program, they will stop the study and open the program to all eligible children.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 3 months and 18 years,
* have at least three chronic medical conditions requiring active management
* were hospitalized or had an emergency department (ED) visit at SCH within the last year
* their PCP is enrolled in the study

Exclusion Criteria:

* had 2+ visits to Pulmonary, Craniofacial, or Rheumatology within the last year
* had 3+ visits to Nephrology, Gastroenterology and has either Short Gut Syndrome or Crohn's Disease, Endocrinology or Neuromuscular Clinic within the last year
* has had 2+ visits to the Neurodevelopmental clinic and is followed by a NDV doctor
* cancer patient
* transplant recipient
* has cystic fibrosis, muscular dystrophy or sickle cell anemia
* has Down Syndrome and does not have any other medical issues aside from developmental delays
* renal patient on dialysis
* had a hospitalization for > 27 days

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 331 (Actual)
Dates: Start 2010-10; Primary Completion 2014-09 (Actual); Study Completion 2017-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita Mangione-Smith, MD, MPH, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Comprehensive Care Management Service
Started | 150 | 181
Completed | 144 | 138
Not Completed | 6 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Comprehensive Care Management Service | Total
Number analyzed (Participants) | 150 | 181 | 331
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 150 | 181 | 331
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (4.8) | 7.9 (5.0) | 8.2 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 92 | 163
  Male | 79 | 89 | 168
Region of Enrollment [Number; unit: participants]
  United States | 150 | 181 | 331

OUTCOME MEASURES:

1. Primary Outcome: Cost of Care
Description: The investigators will examine whether the children in the CCM group experience decreased annual costs of care.
Time Frame: Baseline, 12 month, 18 month
Measure: Mean (95% Confidence Interval); unit: US Dollars
Arm/Group | Control | Comprehensive Care Management Service
Number analyzed (Participants) | 150 | 181
US Dollars
  Health Plan Costs Baseline | 71692 [54511 to 103212] | 70618 [57858 to 95562]
  Health Plan Costs12 month | 37,677 [25811 to 55276] | 56702 [44691 to 80881]
  Health Plan Costs 18 month | 36012 [22888 to 51702] | 52955 [40932 to 74077]

2. Primary Outcome: Health Care Quality Ranking
Description: For Healthcare Quality Rating, the construct is Parent Satisfaction. Parents were asked to rate the quality of the health care their child received. Overall range is 0-100. Higher values equal a better outcome or more satisfaction. Sub scales are not combined. The scale is considered continuous.
Time Frame: Baseline, 12-months, 18-months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Control | Comprehensive Care Management Service
Number analyzed (Participants) | 150 | 181
units on a scale
  Baseline | 79.6 [76.9 to 82.4] | 81.9 [79.4 to 84.4]
  12-Month | 80.9 [78.0 to 83.9] | 88.6 [85.7 to 91.4]
  18-Month | 81.4 [78.2 to 84.6] | 88.2 [85.0 to 91.3]

3. Primary Outcome: ED Visits Per Child
Time Frame: Baseline, 12-month, 18-month
Measure: Mean (95% Confidence Interval); unit: ED visits
Arm/Group | Control | Comprehensive Care Management Service
Number analyzed (Participants) | 150 | 181
ED visits
  Baseline | 0.28 [0.20 to 0.40] | 0.32 [0.24 to 0.43]
  12-Month | .20 [0.14 to 0.29] | .29 [.21 to .40]
  18-Month | .19 [.13 to .27] | .25 [.18 to .34]

4. Primary Outcome: Inpatient Admissions Per Child
Time Frame: Baseline, 12 month, 18 month
Measure: Mean (95% Confidence Interval); unit: admissions per child
Arm/Group | Control | Comprehensive Care Management Service
Number analyzed (Participants) | 150 | 181
admissions per child
  Baseline | .57 [.43 to .74] | .70 [.56 to .88]
  12-Month | .38 [.28 to .51] | .51 [.40 to .65]
  18-Month | .28 [.21 to .39] | .31 [.23 to .41]

5. Primary Outcome: Hospital Days Per Child
Description: Number of days each participant stayed in the hospital; assessed from hospital administrative discharge data
Time Frame: Baseline, 12-Month, 18-Month
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Control | Comprehensive Care Management Service
Number analyzed (Participants) | 150 | 181
days
  Baseline | 1.21 [.86 to 1.74] | 1.34 [.98 to 1.81]
  12-Month | .49 [.34 to .70] | .84 [.61 to 1.14]
  18-Month | .33 [.23 to .47] | .50 [.37 to .69]

6. Secondary Outcome: Physician Satisfaction
Description: Primary care provider (PCP)'s satisfaction with the care coordination program was measured on a scale of 0-100, where the higher number indicates more satisfaction. This variable was collected at baseline and 12-months but was dropped from the 18 month follow-up as previous analysis suggested it was not relevant to the stated objective.
Time Frame: Baseline, 12 Months, 18 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Comprehensive Care Management Service
Number analyzed (Participants) | 150 | 181
units on a scale
  Baseline | 69 (14) | 67 (16)
  12-Month | 71 (13) | 70 (13)

ADVERSE EVENTS:
Arm/Group | Control | Comprehensive Care Management Service
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/181
Other Adverse Events (participants affected / at risk) | 0/150 | 0/181

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes